CLINICAL TRIAL: NCT05977946
Title: Delivering Transcutaneous Auricular Neurostimulation to Regulate Platelet Activity in Healthy Human Subjects
Acronym: HHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spark Biomedical, Inc. (Industry)
Collaborators: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 5L-BLD-03; 23-0265 (Other: Northwell Health)
Record Dates: First submitted 2023-07-14; First posted 2023-08-07 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Hemostasis; Blood Biomarkers
Keywords: Transcutaneous auricular neurostimulation; Transcutaneous auricular vagus nerve stimulation; Blood biomarkers; Neurostimulation; Healthy human

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two 30-minute stimulation sessions. One session will be active and the other sham. Participants are blinded to treatment group as well as the stimulation session.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) (Experimental)
  Interventions: Device: Volta System
- Transcutaneous Auricular Neurostimulation (tAN) (Experimental)
  Interventions: Device: Volta System

INTERVENTIONS:
Device: Volta System — The Volta System is a wearable, battery-operated, neurostimulation system designed to deliver tAN or taVNS. The device will be used to deliver two 30-minute sessions of active or sham therapy according to the participant's randomization group (taVNS or tAN).

SUMMARY:
This study is designed as a randomized, double-blind, sham-controlled, single-center research study in which healthy adults will be randomized 1:1 into one of two experimental groups, to receive transcutaneous auricular vagus nerve stimulation (taVNS) targeting either the auricular branch of the vagus nerve (ABVN) or tAN, which targets the ABVN and the auriculotemporal nerve (ATN):

1. Group 1: Sham taVNS followed by active taVNS
2. Group 2: Sham tAN followed by active tAN

Participants will receive 30 minutes of sham stimulation (taVNS or tAN), followed by active stimulation (taVNS or tAN). Blood biomarkers (local and systemic) will be measured before and at several timepoints after stimulation to measure the molecular and cellular effects of the device.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is between 18 and 65 years of age
2. Participant is English proficient
3. Participant is able to provide informed consent and function at an intellectual level sufficient for study requirements

Exclusion Criteria:

1. Participant has a history of thrombocytopenia (platelet count <100k)
2. Participant has reported coagulopathy (elevated prothrombin time (PT), elevated partial thromboplastin time (PTT), elevated activated clotting time (ACT))
3. Participant has internal bleeding, external bleeding, easy bruising
4. Participant has a history of abnormal bleeding or blood disorder, including anemia or anemia-related disorders
5. Participant has a history of coagulopathy, including hemophilia, stroke, pulmonary embolism, myocardial infarction, or deep vein thromboses
6. Participant has a history of conditions that can cause coagulopathic conditions, including atrial fibrillation, heart valve surgery or replacement, hip or knee replacement, or clotting disorders
7. Participants using coagulation- or platelet-modifying therapies such as clotting factor products, emicizumab, desmopressin acetate, epsilon amino caproic acid, heparin and its derivatives, argatroban, desirudin, bivalirudin, warfarin, dabigatran, apixaban, edoxaban, betrixaban, or aspirin
8. Participant has a history of chronic tobacco use or has ingested nicotine via smoking, vaping, smokeless tobacco, or nicotine patches in the past three months
9. Participant has consumed caffeine within the past 12 hours
10. Participant has received a blood transfusion within 30 days prior to study
11. Participant has a history of epileptic seizures
12. Participant has a history of neurologic diseases or traumatic brain injury
13. Participant has presence of devices (e.g., pacemakers, cochlear prostheses, neurostimulators)
14. Participant has abnormal ear anatomy or ear infection present
15. Women of childbearing potential, not using adequate contraception as per investigator judgment or not willing to comply with contraception for the duration of the study
16. Females who are pregnant, lactating or menstruating
17. Participant has any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants are risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Biomarker of hemostasis (tissue anti-thrombin (TAT) complex) in blood shed from fingerstick | From collection up to 240 minutes, assessed upon receipt of assay results (up to one month)
  Mean TAT levels in shed blood after active stimulation versus sham stimulation within each group
Biomarker of hemostasis (tissue anti-thrombin (TAT) complex) in blood shed from fingerstick | From collection up to 240 minutes, assessed upon receipt of assay results (up to one month)
  Percent change in TAT levels in shed blood after active stimulation between groups (taVNS vs tAN)
Biomarkers of hemostasis (TAT complex, D-dimer, viscoelasticity, coagulation tests (prothrombin time (PT), partial thromboplastin time (PTT)) in circulating blood | From collection up to 240 minutes, assessed upon receipt of assay results (up to one month)
  Mean coagulation biomarker levels in circulating blood after active stimulation versus sham stimulation within each group
Biomarkers of hemostasis (TAT complex, D-dimer, viscoelasticity, coagulation tests (prothrombin time (PT), partial thromboplastin time (PTT)) in circulating blood | From collection up to 240 minutes, assessed upon receipt of assay results (up to one month)
  Percent change in coagulation biomarker levels in circulating blood after active stimulation between groups ( taVNS vs tAN)
Biomarkers of inflammation (tumor necrosis factor (TNF), and interleukin (IL)-1B and IL-6) in circulating whole blood stimulated ex vivo with lipopolysaccharide (LPS) | From collection up to 240 minutes, assessed upon receipt of assay results (up to one month)
  Mean inflammation biomarker levels in LPS-stimulated whole blood after active stimulation versus sham stimulation within each group
Biomarkers of inflammation (tumor necrosis factor (TNF), and interleukin (IL)-1B and IL-6) in circulating whole blood stimulated ex vivo with lipopolysaccharide (LPS) | From collection up to 240 minutes, assessed upon receipt of assay results (up to one month)
  Percent change in inflammation biomarker levels in LPS-stimulated whole blood after active stimulation between groups (taVNS vs tAN)

CONTACTS AND LOCATIONS:
Locations (1):
- The Feinstein Institutes for Medical Research, Manhasset, New York, United States